CLINICAL TRIAL: NCT01112748
Title: Evaluation of Predictors of Response for the Efficacy of Topical Lidocaine Patch (Versatis) on Chronic Neuropathic Pain After Peripheral Nerve Injury
Brief Title: Topical Lidocaine: Predictors of Response in Peripheral Nerve Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Danish Pain Research Center (Other)
Collaborators: Grünenthal Denmark ApS (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIDO-2009
Record Dates: First submitted 2010-04-27; First posted 2010-04-28 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Neuropathic Pain
Keywords: Focal neuropathic pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Topical lidocaine patch — Topical lidocaine patch 5%; up to 3 patches to cover the area of maximum pain for 12 h a day.
  Other Names: Versatis 5% Medicated Plaster, PL21727/0016.

SUMMARY:
The primary purpose is to study the predictive value of preserved nociceptors and large afferent fibers and dynamic mechanical allodynia on the effect of lidocaine patch. The primary outcome measure is the predictive role for these three measures for obtaining a response to lidocaine. A responder is defined as a person with at least a 2-point pain reduction to lidocaine (change in median pain intensity (measured on a 10 point numeric rating scale) of pain from the baseline week to the last week of lidocaine treatment). Secondary effect variable will be efficacy of lidocaine on pain reduction (baseline week versus last week of each treatment) and pain relief (complete, good, moderate, slight, none, or worse) for spontaneous and evoked pain, and effect on ongoing pain, brush evoked allodynia, cold and warm allodynia, and pinprick hyperalgesia evaluated on each visit.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 or more with neuropathic pain after a peripheral nerve injury with a pain intensity of at least 4 on a 0-10 point numeric rating scale.

Exclusion Criteria:

* pregnancy or lactation,
* allergy to lidocaine,
* alcohol abuse,
* psychiatric disorders,
* skin diseases in the area where the patches are to be applied,
* treatment with class I antiarrhythmic agents,
* any treatment within the past one month or concomitantly with Na2+-channel blockers (e.g., mexiletine, phenytoine, propafenone),
* any topical treatment with capsaicin within the last three months before entering the study, or any other topical treatment in the area of neuropathic pain,
* concomitant therapy with TENS or acupuncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity (measured daily on a 10 point NRS)of spontaneous pain from baseline week to last week of treatment | 4 or 12 weeks
  The primary purpose is to study the predictive value of preserved nociceptors and large afferent fibers and dynamic mechanical allodynia on the effect of lidocaine patch. The primary outcome measure is the predictive role for these three measures for obtaining a response to lidocaine. A responder is defined as a person with at least a 2-point pain reduction to lidocaine (change in median pain intensity (measured on a 10 point NRS) of pain from the baseline week to the last week.

SECONDARY OUTCOMES:
Pain relief (complete, good, moderate, slight, none, or worse) for spontaneous and evoked pain | 4 or 12 weeks
Effect on ongoing pain, brush-evoked allodynia, cold and warm allodynia, and pinprick hyperalgesia | 4 or 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nanna B. Finnerup, MD, DMSc., Principal Investigator — Danish Pain Research Center
Locations (1):
- Danish Pain Research Center, Aarhus C, Denmark